CLINICAL TRIAL: NCT01399411
Title: Agricultural Health Study: Health Followup
Brief Title: Agricultural Health Study Follow-up
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911196; 11-E-N196
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-09-16

CONDITIONS: Asthma; Parkinson's Disease
Keywords: Self-Reported; Farming; Agriculture; Disease Validation; Autoimmune Disorders; Natural History
MeSH Terms: conditions — Asthma; Parkinson Disease; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AHS Cohort: licensed pesticide applicators and their spouses from Iowa and North Carolina already enrolled in the Agricultural Health Study (AHS)

SUMMARY:
Background:

- The Agricultural Health Study (AHS) is looking at the long-term health effects of farming exposures including pesticides, crops, and animals. The chronic health effects of exposure to pesticides are easier to study in farmers and their spouses. They know what chemicals they use and tend to live in the same place for most of their adult lives. AHS participants are expected to report any changes in their health. This includes any new medical conditions. Researchers want to follow up on these reports to confirm their accuracy.

Objectives:

- To follow up AHS participants who have self-reported that they have a new disease and confirm their diagnosis.

Eligibility:

- Current AHS participants.

Design:

* Researchers will confirm self-reported changes in medical conditions by contacting the AHS participant to ask for more information.
* The AHS participant will give permission for researchers to contact their doctor to look at their medical records. They will also be asked to provide a cheek swab or saliva sample.
* Diseases of interest are rheumatoid arthritis, lupus, and Sjogren s Syndrome. Other diseases will be followed up in the future. Other diseases will be followed up in the future.

DETAILED DESCRIPTION:
Pesticides are a common environmental exposure due to their widespread use for agricultural, residential, and public health purposes. Farmers and their families represent a unique population for studying the chronic health effects of pesticides because farmers know what chemicals they use, furthermore, farmers tend to remain at the same location over most of their adult life. The Agricultural Health Study (AHS), a cohort of approximately 89,000 pesticide applicators and spouses from Iowa and North Carolina, is the largest US cohort study of individuals working with pesticides. The AHS cohort was enrolled in 1993 to 1997 to assess human health effects associated with well-characterized exposures to pesticides and other agricultural factors. Detailed exposure data were collected at enrollment and in two five-year follow-up interviews. As a result, the AHS has a wealth of information on pesticide use by both farmers and their spouses, as well as the ability to account for changes in pesticide use over time. Information on medical history and important covariates was also collected at enrollment and in the follow-up interviews, and will continue to be collected over time.Only mortality and cancer incidence are updated annually through linkage to vital statistics and cancer registries; all other health outcomes are based on self-reported information from participants.The accuracy of self-reported health outcome information can vary from quite good (e.g., asthma) to poor (e.g., rheumatoid arthritis). In order to ensure high quality epidemiologic analyses, validation of self-reported disease is necessary prior to statistical analysis. To date, several health endpoints have been validated through follow-up with AHS participants and their physicians. The purpose of the current protocol is three-fold: 1) update information on medical history and other important covariates through ongoing follow-up interviews of the cohort; 2) validate self-reported diseases among cohort participants over the duration of cohort follow-up (at least through 2020); and 3) complete initial contact of potential participants to inform them of other health outcome studies being conducted within the cohort by an outside institution.

We will contact AHS cohort members to complete a follow-up interview allowing one of three modes of response: self-administered paper questionnaire, self-administered web survey (CAWI), and interviewer-administered telephone interview (CATI). We will contact proxy respondents if the participant is unable to provide information.

We will validate a variety of diseases of interest as they are ascertained in the cohort. While the characteristics of the diseases may vary, the strategy for disease validation is similar to the cohort wide follow-up. Validation efforts may also include a request for permission to contact the participant s physician, and contacting the physician s office to obtain the relevant medical information. We will contact proxy respondents if the participant is unable to provide information.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

All members of the AHS cohort who were eligible for the Phase 3 interview were eligible for the Phase 4 health follow-up. We will apply the same eligibility criteria for future cohort-wide follow-ups. Individuals who only completed the enrollment questionnaire were excluded from Phase 3 eligibility. Depending upon the disease outcome of interest, we may conduct the disease confirmation and validation efforts under this protocol among all participants in the AHS who provided self-reported diagnoses at any interview (e.g. Baseline, or Phases 2-4). For individuals who are unable to participate, we will allow a proxy to provide the information.

For the validation efforts, individuals who do not confirm their diagnosis of interest (via self or proxy report) will not be asked to provide physician contact for medical records. For specimen collection, we will ask the proxy respondent about whether the individual would be able to provide a sample. In order to obtain MRR we will allow the participant or their medical proxy to sign the form. For cases who are cognitively impaired or deceased, a medical proxy will be identified.

Determination of cognitive impairment will be made by report of proxy or by interviewer during conversation with participant. Because the AHS enrolled husband - wife pairs, we should be able to identify an appropriate proxy for most participants.

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current Agricultural Health Study (AHS) participants (licensed pesticide applicators and their spouses from Iowa and North Carolina)
Sampling Method: Non-Probability Sample
Enrollment: 89656 (Actual)
Dates: Start 2011-07-05 (Actual)

PRIMARY OUTCOMES:
The purpose of the current protocol is three-fold: 1) update information on medical history and other important covariates through ongoing follow-up interviews of the cohort; 2) validate self-reported diseases among cohort participants over the ... | Various phases of follow-up; diseases are validated as they are ascertained
  Changes in health over time.

CONTACTS AND LOCATIONS:
Overall Officials: Dale P Sandler, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Illinois
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina
  - Batelle, Inc., Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided